CLINICAL TRIAL: NCT05336968
Title: Triamcinolone Ketorolac (TriKe) Knee Trial Evaluating the Effectiveness and Possible Superiority of Ketorolac vs. Cortisone When Injected Intra-Articular in Subjects With Osteoarthrosis
Brief Title: Triamcinolone Ketorolac (TriKe) Knee Trial
Acronym: TriKe
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: United Health Services Hospitals, Inc. (Other)
Responsible Party: Principal Investigator, Stanley Hunter, Director, UHSH Concussion Center, United Health Services Hospitals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHSH-9940
Record Dates: First submitted 2022-02-07; First posted 2022-04-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Subjects will receive either ketorolac 30 mg, triamcinolone 40 mg, or a combination of the two medications as a one-time injection into one or both affected knee joint/s.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All staff working with the study subjects will be blinded. Once the subject signs consent, an unblinded study doctor will, using a special method, draw up the appropriate medication and blind the syringe so the the staff giving the medication will not know what is being given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Triamcinolone acetonide - Ropivacaine - Normal Saline (Active Comparator): Subject would receive:
  Triamcinolone acetonide, 40 mg/mL. 1 mL Ropivacaine 0.2%, 2 mL Saline 0.9% 1 mL for a total of 4 mL injected intraarticularly into affected knee/s at randomization
  Interventions: Drug: Triamcinolone acetonide-Ketorolac-Ropivacaine
- Ketorolac - Ropivacaine - Normal Saline (Experimental): Subject would receive:
  Ketorolac 30 mg/mL, 1 mL Ropivacaine 0.2%, 2 mL Saline 0.9% 1 mL for a total of 4 mL injected intraarticularly into affected knee/s at randomization
  Interventions: Drug: Triamcinolone acetonide-Ketorolac-Ropivacaine
- Triamcinolone acetonide - Ketorolac - Ropivacaine (Experimental): Subject would receive:
  Triamcinolone acetonide, 40 mg/mL Ketorolac 30 mg/mL, 1 mL Ropivacaine 0.2%, 2 mL for a total of 4 mL injected intraarticularly into affected knee/s at randomization
  Interventions: Drug: Triamcinolone acetonide-Ketorolac-Ropivacaine

INTERVENTIONS:
Drug: Triamcinolone acetonide-Ketorolac-Ropivacaine — Experimental for Osteoarthrosis of the Knee. One randomized injection to intraarticularly into affected knee at time of randomization

SUMMARY:
Cortisone injections are commonly used in the treatment of osteoarthrosis of the knee, but there are known detriments to cortisone including localized tissue atrophy near the injection site and acceleration of joint degeneration, as well as contraindications, such as uncontrolled diabetes. Ketorolac is a non-steroidal anti-inflammatory with decades of clinical data that is most commonly injected intramuscularly. There is rising interest in using ketorolac as an intra-articular injectant substitute or adjunctive to cortisone. This may potentially improve clinical outcomes or decrease adverse effects. Although intra-articular use of ketorolac is increasing in orthopedics and sports medicine, there is limited data in the literature comparing these two injectants in prospective, randomized trials, and no data that evaluates combining the two injectants. Primary objectives are to evaluate the efficacy of intra-articular ketorolac compared to cortisone on knee osteoarthrosis and to evaluate whether the combination of ketorolac and cortisone is superior to either alone.

DETAILED DESCRIPTION:
Charts will be prescreened for diagnosis or suspicion of osteoarthritis of the knee by the study staff. Those charts identified will be flagged for possible inclusion in the study. The receptionist will give the prospective subject a copy of the consent to read while they are in the waiting room. Once they are taken back to the room, the investigator will review the study with them. If they are agreeable, they will sign the consent and a copy will be given to them and a copy will be scanned into the Electronic Medical Record (EMR). The investigator will then notify the unblinded investigator, who will randomize the subject and prepare the medication in a blinded fashion. The subject will receive either ketorolac 30 mg, triamcinolone 40 mg, or a combination of the two medications as a one-time injection into the affected knee joint/s. The subject will be asked to complete a survey prior to receiving the injection, and again at 1 week, 6 weeks, and 12 weeks post injection. If necessary, an additional survey will be completed at 24 weeks post injection.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain with diagnosis of osteoarthritis/osteoarthrosis
* Weight-bearing x-rays within the last year adequate to assess Kellgran-Lawrence OA stage
* Age > 21
* English proficiency sufficient to complete surveys
* Willing to complete follow-up surveys

Exclusion Criteria:

* Prior knee injection in last 3 months
* Knee surgery within the last year
* Contraindications to Cortisone, Ketorolac, or local anesthetic
* Uncontrolled diabetes
* Systemic steroid use in last 3 months
* BMI > 50
* Non-ambulatory
* Known kidney disease
* Current opioid use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported outcomes as measured by Modified KOOS scores | 12 -24 weeks
  Change in patient reported outcomes as measured by Modified Knee Injury and Osteoarthritis Outcome Score (KOOS, higher is better [0-100]).
Evaluate whether the combination of ketorolac and cortisone is superior to either alone as measured by Modified KOOS | 12 -24 weeks
  Change in patient reported outcomes as measured by Modified Knee Injury and Osteoarthritis Outcome Score (KOOS, higher is better [0-100])

SECONDARY OUTCOMES:
Change in patient reported outcomes as measured by VAS | 12 -24 weeks
  Change in patient reported outcomes as measured by Visual Analog Scale (VAS, lower is better [0-100])
Evaluate whether the combination of ketorolac and cortisone is superior to either alone as measured by VAS | 12 -24 weeks
  Change in patient report outcomes as measured by Visual Analog Scale (VAS, lower is better [0-100])

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hunter, MD, Principal Investigator — United Health Services Hospitals, Inc.
Locations (1):
- United Health Services Sports Medicine Department, Vestal, New York, United States